CLINICAL TRIAL: NCT02362048
Title: A Phase 2 Proof-of-Concept Study of ACP-196 Alone and in Combination With Pembrolizumab in Subjects With Advanced or Metastatic Pancreatic Cancer
Brief Title: ACP-196 Alone and in Combination With Pembrolizumab in Subjects With Advanced or Metastatic Pancreatic Cancer
Acronym: KEYNOTE144
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE-ST-003
Record Dates: First submitted 2015-01-28; First posted 2015-02-12 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — acalabrutinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: Arm 1 (Experimental): ACP-196 alone
  Interventions: Drug: ACP-196
- Experimental: Arm 2 (Experimental): ACP-196 in combination with pembrolizumab
  Interventions: Drug: ACP-196 in combination with pembrolizumab

INTERVENTIONS:
Drug: ACP-196
  Arms: Experimental: Arm 1
Drug: ACP-196 in combination with pembrolizumab
  Arms: Experimental: Arm 2

SUMMARY:
ACP-196 Alone and in Combination with Pembrolizumab in Subjects with Advanced or Metastatic Pancreatic Cancer

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age
* ECOG performance status of 0 or 1
* Histologically or cytologically confirmed advanced pancreatic ductal adenocarcinoma that is unresectable or metastatic
* Prior therapy with ≥ 1 systemic chemotherapy regimen for unresectable or metastatic pancreatic cancer or unwilling/unable to receive systemic chemotherapy

Exclusion Criteria:

* Prior malignancy (other than pancreatic cancer), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for ≥ 2 years or which will not limit survival to < 2 years.
* Known central nervous system (CNS) metastases and/or carcinomatous meningitis
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease, partial or complete bowel obstruction
* Breastfeeding or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Acerta Clinical Trial, Study Director — 1-888-292-9613; acertamc@dlss.com
Locations (1):
- Houston, Texas, United States

REFERENCES:
- [Derived] Overman M, Javle M, Davis RE, Vats P, Kumar-Sinha C, Xiao L, Mettu NB, Parra ER, Benson AB, Lopez CD, Munugalavadla V, Patel P, Tao L, Neelapu S, Maitra A. Randomized phase II study of the Bruton tyrosine kinase inhibitor acalabrutinib, alone or with pembrolizumab in patients with advanced pancreatic cancer. J Immunother Cancer. 2020 Feb;8(1):e000587. doi: 10.1136/jitc-2020-000587. PMID 32114502

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 - Acalabrutinib Monotherapy: Acalabrutinib 100 mg administered orally (PO) twice daily (BID)
- Arm 2- Acalabrutinib+Pembrolizumab: Acalabrutinib 100 mg PO BID plus pembrolizumab 200 mg administered as an intravenous (IV) infusion every 3 weeks (Q3W)
Period: Overall Study
Arm/Group | Arm 1 - Acalabrutinib Monotherapy | Arm 2- Acalabrutinib+Pembrolizumab
Started | 37 (37 enrolled but only 35 received study medication.) | 40 (40 enrolled but only 38 received study medication.)
Enrolled | 37 | 40
Received Study Medication | 35 | 38
Discontinued Study | 37 | 40
Completed | 0 | 0
Not Completed | 37 | 40

BASELINE CHARACTERISTICS:
Groups:
- Monotherapy Arm: ACP-196 alone
  ACP-196
- Combination Arm: ACP-196 in combination with pembrolizumab
  ACP-196 in combination with pembrolizumab
- Total: Total of all reporting groups
Arm/Group | Monotherapy Arm | Combination Arm | Total
Number analyzed (Participants) | 35 | 38 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 23 | 43
  >=65 years | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: Year] | 62.9 (8.19) | 61.3 (10.94) | 62.1 (9.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 17 | 19 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 34 | 33 | 67
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 29 | 33 | 62
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 35 | 38 | 73

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response Advanced or Metastatic Pancreatic Cancer.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Every 12 weeks for up to 2 years.
Population: All participants with Baseline and at least one post-baseline target lesion measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Acalabrutinib Monotherapy | Arm 2- Acalabrutinib+Pembrolizumab
Number analyzed (Participants) | 29 | 27
Participants | 0 | 3

ADVERSE EVENTS:
Time Frame: AE collected time frame was From the date of the first dose of study drug, through the treatment phase, and within 30 days following the last dose of Acalabrutinib or within 90 days following the last dose of Pembrolizumab.
Description: Subjects with multiple events for a given preferred term (PT) were counted only once for each PT. If the same event term was reported more than once for a subject, only the event with the highest grade was included.
Arm/Group | Arm 1 - Acalabrutinib Monotherapy | Arm 2- Acalabrutinib+Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 30/35 | 34/38
Serious Adverse Events (participants affected / at risk) | 14/35 | 26/38
Other Adverse Events (participants affected / at risk) | 34/35 | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Acalabrutinib Monotherapy (N=35) | Arm 2- Acalabrutinib+Pembrolizumab (N=38)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 5
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdomincal Distension (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 0
Upper Gastrointestinal Haemorrage (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 2
Autoimmune Hepatitis (Hepatobiliary disorders) | 0 | 1
Bile Duct Obstruction (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 0
Portal Vien Thrombosis (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 1 | 1
Abdominal Infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0
Escherichia Sepsis (Infections and infestations) | 1 | 0
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 1
Hepatic Infection (Infections and infestations) | 1 | 0
Klebsiella Sepsis (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Blood Bilirubin Increased (Investigations) | 0 | 1
Troponin T Increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Failure to Thrive (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant Ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Cerebellar Infarction (Nervous system disorders) | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Malignant Bowel Obstruction (Gastrointestinal disorders) | 0 | 1
Oesophagitis Ulcerative (Gastrointestinal disorders) | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Acalabrutinib Monotherapy (N=35) | Arm 2- Acalabrutinib+Pembrolizumab (N=38)
Anaemia (Blood and lymphatic system disorders) | 12 | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4
Sinus Tachycardia (Cardiac disorders) | 2 | 1
Abdominal Pain (Gastrointestinal disorders) | 10 | 21
Nausea (Gastrointestinal disorders) | 8 | 14
Constipation (Gastrointestinal disorders) | 8 | 13
Vomiting (Gastrointestinal disorders) | 6 | 15
Abdominal Distension (Gastrointestinal disorders) | 5 | 9
Fatigue (General disorders) | 11 | 16
Oedema Peripheral (General disorders) | 9 | 5
Pyrexia (General disorders) | 5 | 9 — General Disorders and Administration Site Conditions
Chills (General disorders) | 2 | 4
Asthena (General disorders) | 3 | 2 — General Disorders and Administration Site Conditions
Pain (General disorders) | 1 | 2 — General Disorders and Administration Site Conditions
Influenza like Illness (General disorders) | 1 | 2 — General Disorders and Administration Site Conditions
Chest Discomfort (General disorders) | 0 | 2 — General Disorders and Administration Site Conditions
Chest Pain (General disorders) | 0 | 2 — General Disorders and Administration Site Conditions
Mucosal Inflammation (General disorders) | 0 | 2 — General Disorders and Administration Site Conditions
Urinary Tract Infection (Infections and infestations) | 2 | 5
Pneumonia (Infections and infestations) | 1 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 2
Blood Alkaline Phosphatase Increased (Investigations) | 2 | 6
Blood Creatinine Increased (Investigations) | 5 | 4
Alanine Aminotransferase Increased (Investigations) | 3 | 5
Blood Bilirubin Increased (Investigations) | 1 | 4
Aspartate Aminotransferase Increased (Investigations) | 2 | 4
Platelet Count Decreased (Investigations) | 5 | 1
Lymphocyte Count Decreased (Investigations) | 0 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 11 | 18
Dehydration (Metabolism and nutrition disorders) | 6 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 8 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 11 | 11
Dizziness (Nervous system disorders) | 4 | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 3 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 7
Dry Skin (Skin and subcutaneous tissue disorders) | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 4
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 2
Hypotension (Vascular disorders) | 4 | 5
Ascites (Gastrointestinal disorders) | 4 | 9
Diarrhoea (Gastrointestinal disorders) | 6 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 3
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 6
Anxiety (Psychiatric disorders) | 3 | 3
Depression (Psychiatric disorders) | 1 | 2
Acute Kidney Injury (Renal and urinary disorders) | 2 | 3
Haematuria (Renal and urinary disorders) | 2 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Stomatitis (Gastrointestinal disorders) | 2 | 1
Weight Decreased (Investigations) | 4 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 3
Tachycardia (Cardiac disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 4
Candida Infection (Infections and infestations) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/48/NCT02362048/SAP_000.pdf
  • Study Protocol (2016-01-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT02362048/Prot_001.pdf